CLINICAL TRIAL: NCT06749314
Title: Comparison of Endoscopic Lumbar Decompression and Minimal Invasive Surgery Transforaminal Lumbar Interbody Fusion (MIS-TLIF) for Degenerative Lumbar Spondylolisthesis: A Randomized Controlled Study
Brief Title: Comparison of Endoscopic Lumbar Decompression and Minimally Invasive Transforaminal Lumbar Interbody Fusion(MIS-TLIF) for Degenerative Lumbar Spondylolisthesis
Acronym: MIS-TLIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 024/2567
Record Dates: First submitted 2024-11-04; First posted 2024-12-27 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Lumbar Spondylolisthesis; Lumbar Degenerative Disease; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: The participants were randomized into two group with computer generated block-of-four randomization with allocation 1:1 into two groups. The control group recieved MIS TLIF while the experimental group recieved endoscopic decompression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar Endoscopic - Unilateral Laminotomy for Bilateral Decompression (Experimental): using endoscopic decompression for treatment
  Interventions: Procedure: Lumbar Endoscopic - Unilateral Laminotomy for Bilateral Decompression
- MIS-TLIF: Minimal Invasive Surgery - Transforaminal Lumbar interbody Fusion (No Intervention): Using conventional treatment, minimal invasive decompression with interbody fusion surgery for treatment in control groups

INTERVENTIONS:
Procedure: Lumbar Endoscopic - Unilateral Laminotomy for Bilateral Decompression — The LE-ULBD: Lumbar Endoscopic - Unilateral Laminotomy for Bilateral Decompression is a single portal through lamina with instrument to decompression both side of the spinal canal, giving strength of preserve facet joint, preserve spinal musculature, mitigate the risk of adjacent fusion and lesser bleeding
  Other Names: LE-ULBD; endoscopic decompression
  Arms: Lumbar Endoscopic - Unilateral Laminotomy for Bilateral Decompression

SUMMARY:
Comparing the functional and radiographic outcomes in surgical treatment in failed conservative treatment, single-level low grade degenerative lumbar spondylolisthesis between Minimal Invasive Surgery Transforaminal Lumbar Interbody Fusion, which is conventional treatment recently, and Endoscopic Lumbar Decompression, which is minimal invasive in symptomatic treatment.

DETAILED DESCRIPTION:
This was a randomized controlled trial in patient with single-level low grade degenerative lumbar spondylolisthesis with failed conservatives treatment, by comparing two group of surgical intervention between Minimally Invasive Transforaminal Lumbar Interbody Fusion (MIS TLIF) and Endoscopic lumbar decompression using functional outcomes.

The participants were randomized into two groups with 33 cases each group (Total = 66) by using computer generated program with block of four randomization with allocation ratio 1:1. The control group received conventional treatment which is Minimal Invasive Surgery Transforaminal Lumbar Interbody Fusion while the experimental group received endoscopic lumbar decompression. Using ODI score as primary outcome. Data were analyzed using chi-square test for categorical data (eg, sex, symptoms of weakness and numbness, level of spondylolisthesis) and unpaired T-test for continuous data (eg. VAS score, ODI, slippage percentage, lumbar lordosis degree, slip angle, op time) which considered significant difference of the outcomes when p < 0.05 with a power of 80%. Consider endoscopic decompression is non-inferiority to MIS-TLIF when upper limit of the one-sided 95%CI for the differences in ODI means is less than margin (12.8 points) If the results show that endoscopic decompression is non-inferiority to MIS TLIF, endoscopic lumbar decompression may be a choice of treatments giving benefit of minimal invasive surgery and avoid interbody fusion complication such as pseudoarthrosis, adjacent problems and operative blood loss

ELIGIBILITY:
Inclusion Criteria:

* Single level lumbar degenerative spondylolisthesis (Meyerding Grading Grade I or II).
* Failed conservative treatment for at least 3 months.
* No instability evidence of levels of lesion (Consideration from translation more than 5 mm or angulation change more than 10 degree in flexion and extension L-S plain films ).
* Able to follow up for at least 12 months.
* Patient who vorantarily agree to participate in research.

Exclusion Criteria:

* Patients with severe foraminal stenosis diagnosed by MRI.
* Patients who have previously undergone lumbar spine surgery (revision surgery).
* Patients with other abnormalities in the lumbar spine, such as infection, tumors, or fractures.
* Patients who cannot undergo surgery due to underlying conditions or who cannot maintain the prone position for extended periods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index score | 1 year; Preoperative and post-operative at 12 months
  The Oswestry Disability Index (ODI) is a patient-completed questionnaire made up of 10 questions, each with six statements that are scored from 0 to 5. The questions cover a range of activities, including pain intensity, personal care, walking, sleeping, social life, and travel. The ODI score ranges from 0% to 100%, with higher scores indicating more severe disability:
  0-20%: Mild disability 20-40%: Moderate disability 40-60%: Severe disability 60-80%: Disabling 80-100%: Bedridden or functional impairment

SECONDARY OUTCOMES:
Visual analog scale of leg pain | 1 year; Preoperative and post-operative at 1,3,6 and 12 months
  Pain score of leg pain from 1-10 determined by measuring in millimeters from the left hand end of the line to the point that the patient marks
Visual analog scale of back pain | 1 year; Preoperative and post-operative at 1,3,6 and 12 months
  Pain score of back pain from 1-10 determined by measuring in millimeters from the left hand end of the line to the point that the patient marks
Modified Macnab criteria | 1 year; Preoperative and post-operative at 1,3,6 and 12 months
  The Modified MacNab criteria are a set of guidelines used to assess the outcomes of spinal surgery, particularly in evaluating the effectiveness of procedures like discectomy or spinal fusion
Operative time | 1 day; From patient's skin is cut, through each intervention surgery completion (minute) when the skin is closed
  Operative time that using in each intervention start from when patient's skin is cut and stop when it is closed. Measure in minute
Length of hospital stay | 1 year; The date from the patients had been admitted to discharge
  Total days that the patients had been admitted to discharge
Amount of blood loss | 1 day; Start from the skin's is cut through surgery period and postoperative until the drain bottle was removed.
  Total blood loss during surgery and postoperative measuring from visual estimation, gravimetric method, suction bottle and drainage bottle after surgery.
Radiographic outcomes: lumbar slip percentage | 1 year; Preoperative and post-operative at 0,6 and 12 months
  Comparing lumbar slip percentage which calculated by measuring the displacement of the upper vertebral body relative to the lower vertebral body on a lateral radiograph preoperative and postoperative at each time point by:
  1. Draw a line along the posterior border of the lower vertebral body
  2. Draw a line perpendicular to the first line at the top of the lower vertebral body
  3. Draw a line along the posterior border of the upper vertebral body
  4. Calculate the percentage of the anterior translation of the upper vertebral body relative to the width of the lower vertebral body.
Radiographic outcomes: Slip angle | 1 year; Preoperative and post-operative at 0,6,12 months
  The lumbar slip angle in spondylolisthesis is measured by drawing lines on a lateral X-ray and measuring the angle between them:
  1. Extend a line along the anterior border of the upper vertebral body spondylolisthesis level
  2. Draw a line along the posterior border of the lower vertebra spondylolisthesis level
  3. Draw a line perpendicular to the posterior aspect of the first lower vertebra
  3. Measure the angle between the line perpendicular to the first lower vertebra and a line parallel to the inferior end plate of upper vertebra A slip angle greater than 45 degrees is associated with a higher risk of instability, slip progression, and post-op pseudo-arthrosis.
Radiographic outcomes: lumbar lordosis degree | 1 year; Preoperative and post-operative at 0,6,12 months
  The lumbar lordosis angle in spondylolisthesis is measured in degree by drawing lines on an X-ray film and calculating the angle formed by their intersection:
  1. Draw a line tangent to the superior endplate of the first lumbar vertebra (L1)
  2. Draw a line tangent to the inferior endplate of the fifth lumbar vertebra (L5)
  3. Draw a perpendicular line to each tangent
  4. The angle formed by the intersection of the two perpendicular lines is the lumbar lordosis angle

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Nadhana Memorial Hospital, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No